CLINICAL TRIAL: NCT01545141
Title: Randomized Phase 1/2 Evaluation of Neoadjuvant Administration of a Chemokine-Modulatory Regimen in Patients With Recurrent Resectable Colorectal Cancer
Brief Title: Chemokine-Modulatory Regimen for Recurrent Resectable Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-131; 10-131 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: metastatic; recurrent; peritoneal metastasis; cytoreductive surgery; hyperthermic intraperitoneal chemoperfusion; HIPEC; hepatic metastasis; extrahepatic metastasis; vaccine
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Celecoxib; Introns; Interferon alpha-2; Interferon-alpha; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Surgery only (No Intervention): Surgical resection only, performed as standard of care for the disease
- Chemokin Modulatory Regimen (5 MU/m2) (Experimental): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 5 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Interventions: Drug: Chemokin Modulatory Regimen (5 MU/m2)
- Chemokin Modulatory Regimen (10 MU/m2) (Experimental): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 10 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Interventions: Drug: Chemokin Modulatory Regimen (10 MU/m2)
- Chemokin Modulatory Regimen (20 MU/m2) (Experimental): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 20 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Interventions: Drug: Chemokin Modulatory Regimen (20 MU/m2)

INTERVENTIONS:
Drug: Chemokin Modulatory Regimen (5 MU/m2) — Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 5, 10, and 20 MU/m2.
  Other Names: Celebrex; INTRON A; Interferon-alpha 2b; IFN-alpha; Ampligen; rintatolimod
  Arms: Chemokin Modulatory Regimen (5 MU/m2)
Drug: Chemokin Modulatory Regimen (10 MU/m2) — Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery
  Other Names: Celebrex; INTRON A; Interferon-alpha 2b; IFN-alpha; Ampligen; rintatolimod
  Arms: Chemokin Modulatory Regimen (10 MU/m2)
Drug: Chemokin Modulatory Regimen (20 MU/m2) — Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery
  Other Names: Celebrex; INTRON A; Interferon-alpha 2b; IFN-alpha; Ampligen; rintatolimod
  Arms: Chemokin Modulatory Regimen (20 MU/m2)

SUMMARY:
Determine the safety of a combination of IFN, celecoxib, and rintatolimod for patients with recurrent colorectal cancer. This will also test whether the above combination can help the immune system to fight the tumors. The results will allow the investigators to determine the "preferred" combination for subsequent extended studies.

DETAILED DESCRIPTION:
A previously-demonstrated correlation between the density of CRC-infiltrating effector T cells and long-term outcomes (Galon et al., 2006; Pages et al., 2005) has been established. In preclinical ex vivo studies performed using explants of resected metastatic CRC, the combination of IFNα with nonselective or COX2-selective inhibitors of prostaglandin synthesis resulted in elevated production of the effector T cell-attracting chemokines CXCL10 and CCL5. This was associated with concomitant suppression of the intratumoral expression of CCL22, a Treg-attracting chemokine (Muthuswamy et al 2008 Canc Res, and Muthuswamy et al, submitted to Canc Res 2011). However, in a subset of patients, the optimal results, particularly with regard to CCL5 induction, required additional stimulation by a third agent, poly-I:C (a toll-like receptor -TLR Ligand).

Therefore, the investigators seek to establish the safety profile of a novel chemokine regimen consisting of IFN, celecoxib and poly-I:C. The investigators also hypothesize that the proposed neoadjuvant chemokine modulation treatment in recurrent CRC patients undergoing tumor resection may increase the density of tumor infiltrating lymphocytes (TILS).

In addition, treatment in the neoadjuvant setting will allow a comparative analysis of the effect of chemokine modulation on the local recruitment of effector-type T cells and the de-recruitment of Treg within resected tumor tissues; helping to determine the "preferred" chemokine-modulating regimen for subsequent extended studies. Such prospective studies will focus on using combinations of chemokine modulation and cancer vaccines in patients with CRC. The investigators have, for example, recently observed that αDC1, a new type of DC vaccine (Kalinski and Okada, 2010; Mailliard et al., 2004) is particularly effective in inducing the effector pathway of T cells differentiation. This was manifested by the induction of tumor-killing function and the induction of effector-type chemokine receptors (CXCR3 and CCR5) (Kalinski and Okada, 2010; Watchmaker et al., 2010). Combining the αDC1 vaccine to a safe, tolerable and efficacious CKM regimen may hold promise for patients with poor prognostic CRC.

ELIGIBILITY:
Inclusion:

* Recurrent and/or metastatic resectable colorectal cancer, including disease within the abdomen and pelvis with no evidence of extra-abdominal metastases. Isolated resectable pulmonary metastasis are allowable in the absence of intra-abdominal metastasis. Intra-abdominal disease includes: isolated hepatic metastasis/metastases (see next inclusion criteria point), isolated peritoneal metastasis, peritoneal carcinomatosis (including patients undergoing cytoreductive surgery alone or in combination with hyperthermic intraperitoneal chemoperfusion - HIPEC), or a combination of hepatic and extrahepatic metastasis.
* Patients with isolated hepatic metastasis must satisfy a Clinical Risk Score of 3 or higher (see Appendix C)
* Eligible patients are expected to have a complete resection based on preoperative imaging. Any patient not found to be able to have complete resection will not be eligible for this study.
* No chemotherapy, radiotherapy, major surgery, or biologic therapy within 3 weeks of protocol treatment
* An ECOG performance status of 0, 1, or 2.
* Age equal to 18 years or older.
* Must have normal organ and marrow function as defined below:

  * Platelet ≥ 75,000/µL
  * Hemoglobin ≥ 9.0 g/dL
  * Hematocrit ≥ 27.0%
  * Absolute Neutrophil Count (ANC) ≥ 1500/µL
  * Creatinine < institutional upper limit of normal (ULN) OR
  * Creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels greater than ULN
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤ 2.5 X institutional upper limit of normal (ULN)
  * Serum amylase and lipase within normal limits.
* Patient must be able to understand and be willing to sign a written informed consent document.

Exclusion:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment.
* Patients with active autoimmune disease or history of transplantation.
* Patients who are pregnant or nursing. Women of childbearing potential (WOCBP) will have to undergo a urine pregnancy test as part of screening.
* Patients with comorbid medical conditions that render them unfit for surgery.
* Metastatic or recurrent disease that is deemed partially resectable or unresectable based on preoperative imaging.
* Metastatic disease outside the confines of the abdomen, pelvis and thorax (e.g bone, brain)
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
  * Patients with a New York Heart Association classification of III or IV (Appendix A)
* History of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years. Patients with ulceration, bleeding or perforation in the lower bowel are not excluded.
* Prior allergic reaction or hypersensitivity to sulfonamides, celecoxib, or NSAIDs.
* Patients are ineligible if they plan on regular use of NSAIDs at any dose more than 2 times per week (on average) or aspirin at more than 325 mg at least three times per week, on average. Low-dose aspirin not exceeding 100 mg/day is permitted. Patients who agree to stop regular NSAIDs or higher dose aspirin are eligible and no wash out period is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2016-04-08 (Actual); Study Completion 2017-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amer H Zureikat, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 Patients were enrolled in Phase I. 6 Patients were enrolled in Phase II prior to study termination (funding).
Groups:
- Chemokin Modulatory Regimen (5 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 5, 10, and 20 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 5, 10, and 20 MU/m2.
Period: Overall Study
Arm/Group | Surgery Only | Chemokin Modulatory Regimen (5 MU/m2) | Chemokin Modulatory Regimen (10 MU/m2) | Chemokin Modulatory Regimen (20 MU/m2)
Started (9 patients in Phase I. 6 patients randomized in Phase II (2 to surgery alone and 4 to 20 MU/m2)) | 2 | 3 | 3 | 7
Completed | 2 | 3 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 9 patients in Phase I 6 patients in Phase II
Groups:
- Chemokine Modulatory Regimen (5 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 5 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 5 MU/m2.
- Chemokine Modulatory Regimen (10 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 10 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 10 MU/m2.
- Chemokine Modulatory Regimen (20 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 20 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 20 MU/m2.
- Total: Total of all reporting groups
Arm/Group | Surgery Only | Chemokine Modulatory Regimen (5 MU/m2) | Chemokine Modulatory Regimen (10 MU/m2) | Chemokine Modulatory Regimen (20 MU/m2) | Total
Number analyzed (Participants) | 2 | 3 | 3 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 6 | 9
  >=65 years | 1 | 2 | 2 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (4.2) | 62.7 (13.7) | 60.0 (15.9) | 47.1 (15.3) | 55.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 4 | 6
  Male | 2 | 1 | 3 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Tumor-infiltrating CD8+ Cells.
Description: This will be assessed by the increase in the total number of tumor-infiltrating CD8+ T cells in the resected, recurrent CRC lesions (measured as the ratio between the CD8 mRNA message and the expression of the housekeeping gene HPRT), comparing Arm A and Arm B.
Time Frame: Day of surgery: day 8-10
Population: The study was terminated prior to completion of enrollment for Phase II and the T-cell analysis was not completed.
Groups:
- Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 2 dose of 20 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 20 MU/m2.
Arm/Group | Surgery Only | Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Treatment Related Adverse Events
Description: The number of adverse events experienced within 1 week of treatment. This was completed for the Phase II portion of the study.
Time Frame: 1 week
Population: The study was terminated prior to completion of enrollment for Phase II. The Phase II portion of the study involved Surgery alone and Chemokin Modulatory Regimen prior to surgery at 20 MU/m2.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery Only | Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2)
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were measured for 30 days after treatment.
Description: Definitions are as described in clinicaltrials.gov
Groups:
- Chemokin Modulatory Regimen Prior to Surgery (5 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 5 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 5 MU/m2.
- Chemokin Modulatory Regimen Prior to Surgery (10 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 10 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 10 MU/m2.
- Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2): Chemokine Modulatory Regimen monday through Friday prior to surgery:
  400 mg celecoxib for 5 days IFN by intravenous infusion (IV) (Phase 1 dose escalation of 20 MU/m2) for 5 days Rintatolimod 200 mg by IV infusion for 5 days
  Chemokine modulatory regimen: Celecoxib: 200 mg twice/day M-F of the week prior to scheduled surgery rintatolimod: 200 mg i.v. administration M-F of the week prior to scheduled surgery IFN: i.v. administration, M-F of the week prior to scheduled surgery. Dose escalation evaluating 20 MU/m2.
Arm/Group | Surgery Only | Chemokin Modulatory Regimen Prior to Surgery (5 MU/m2) | Chemokin Modulatory Regimen Prior to Surgery (10 MU/m2) | Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 1/3 | 1/7
Other Adverse Events (participants affected / at risk) | 0/2 | 3/3 | 3/3 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Only (N=2) | Chemokin Modulatory Regimen Prior to Surgery (5 MU/m2) (N=3) | Chemokin Modulatory Regimen Prior to Surgery (10 MU/m2) (N=3) | Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2) (N=7)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Only (N=2) | Chemokin Modulatory Regimen Prior to Surgery (5 MU/m2) (N=3) | Chemokin Modulatory Regimen Prior to Surgery (10 MU/m2) (N=3) | Chemokin Modulatory Regimen Prior to Surgery (20 MU/m2) (N=7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 3 (4) | 3 (3) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 3 (4) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No